CLINICAL TRIAL: NCT04299685
Title: What Are the Family Barriers and Facilitators of Healthy Eating Habits Among Adolescents?
Brief Title: Family Factors of Eating Habits Among Adolescents
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, The University of Hong Kong
Other Study IDs: UW20-007
Record Dates: First submitted 2020-03-02; First posted 2020-03-09 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Eating Habit; Healthy Diet
Keywords: Eating habits, barriers, facilitators, adolescents
MeSH Terms: conditions — Feeding Behavior | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Qualitative family interviews of 20 family units, or more until data saturation, of at least one parent and one adolescent (aged 10-19 year old) will be conducted based on deductive thematic approach. Each interview will last for about an hour, be conducted in Cantonese, and audio-taped for transcription in verbatim in Chinese.

SUMMARY:
Healthy eating is a key preventive approach to combat the rising prevalence of non-communicable diseases (NCD) worldwide. The dietary habit established during adolescence has high tendency to continue to adulthood, and is affected by family factors in multiple dimensions. Kerry Group Kuok Foundation (Hong Kong) Limited (KGKF) initiated the Trekkers Family Enhancement Scheme (TFES) in 2012 to empower low-income families in Tung Chung to self-care and development. In response to the persistent unhealthy eating habits among these families despite a series of nutrition workshops incorporating short talks and sharing of healthy recipes, this study aims to investigate the barriers, facilitators and strategies that enable adolescents from low income families to develop a healthy eating habit. Qualitative family interviews of 20 family units, or more until data saturation, of at least one parent and one adolescent (aged 10-19 year old) will be conducted based on deductive thematic approach. Each interview will last for about an hour, be conducted in Cantonese, and audio-taped for transcription in verbatim in Chinese. The data will be coded independently into broad themes in English by two members of the research team. This research can provide an insight into personal and familial factors and potential strategies influencing eating habits of adolescents, which can guide the development of effective interventions to promote healthy eating in low-income families.

DETAILED DESCRIPTION:
Background:

Healthy lifestyle is a key preventive approach to combat the rising prevalence of non-communicable diseases (NCD) worldwide], among which diet is highlighted as a modifiable risk factor of the most common NCD, namely hypertension, diabetes mellitus and coronary heart disease. Adolescence is a transitioning stage from parent-dependence to increasing autonomy in behavior including healthy or risky behavior. The dietary habit established in this period has high tendency to continue to adulthood.

Many national dietary recommendations were established to promote quality diet in order to prevent NCD in the population. They commonly cover starchy foods, vegetables and fruits, protein food, dairy, fats/oils and sugars/sweets. Some guidelines are more generic on certain food groups or overall diet, such as "Eat plenty of cereals, preferably wholegrain, and potatoes" and "Eat foods from each food group every day to have a complete diet". Others provide quantified suggestion, for example, "Consume three or more servings of vegetables and at least two servings of fruit per day" and "Less than 5 g of salt per day and use iodized salt". However, the adherence rate to these recommendations remains low in most other populations, with at least 60% of general population having insufficient intake of fruit and vegetables and overconsumption of added sugar and sodium. The Hong Kong Population Health Survey 2014/15 found that 94.4% of local residents aged 15 or above consumed less than the recommended 5 servings of fruit and vegetables each day, and 21.5% had eaten snacks with high salt content at least once a week in the past one month.

Many studies have explored the contributing factors of eating habits among adolescents. Based on Health Belief Model, they can be categorized into A) socio-psychological variables including familial factors and peer influence; B) cue to action by media, home and school environment; C) perceived benefits on personal health; and D) perceived barriers on personal preference towards food, logistic and lack of motivation. Family factors affect adolescents' eating pattern in multiple dimensions, including parental modeling, home food environment, education on healthy eating and mealtime structure.

The Innocenti Framework on Food System for Children and Adolescents explains the family role in adolescents' diet. The framework was developed by UNICEF in 2018 to address the direct and underlying factors, drivers, and dynamics between food, people, and the planet. It comprises four determinants, namely Food Supply Chain, External Food Environments, Personal Food Environments, and Behaviors of Caregivers, Children and Adolescents. The former two determinants outline the structural factors of the system, such as taxation, advertisement on media, and food availability in the market. The latter two look into the social and personal variables, which comprise individual and household factors. Family factors including accessibility, affordability and convenience of healthy food are personal environment determinants; intra-household dynamics (e.g. care practices, control on household expenses), food preparation, socioeconomic characteristics and eating patterns are behavioral determinants in the family. The framework emphasizes the dynamics between the determinants and diets of children and adolescents. For instance, food price and availability in the market contribute to personal food environments, which is also influenced by personal desirability and food preparation skill. Parental behaviors become a buffer between food environments and children's diets.

Socioeconomic status (SES) has proven positive association with diet quality. Reviews showed that low SES individuals preferred energy-dense, nutrient-poor diets with insufficient whole grains, low-fat foods and fresh produce but high in added sugars or fats. Similar socioeconomic association with dietary pattern was found in adolescents and in Hong Kong. This can be explained by the special challenges that low-income families face: 1) Economic constraint poses food-cost concern where nutritious foods generally cost more and parents prioritize children's preference to avoid food waste. 2) Employed parents usually have long working hours and fail to develop healthy eating behavior with their children. Time pressure also promotes dining-out at fast food shop as alternative to home meal preparation. 3) Low education level may lead to the lack of dietary knowledge for food choice and preparation. 4) The access to the healthy foods is limited by the availability in the community as the families seldom do grocery shopping in distant places.

The Trekkers Family Enhancement Scheme (TFES) was initiated by a philanthropic group, Kerry Group Kuok Foundation (Hong Kong) Limited (KGKF) since 2012. It aims to empower low-income families in Tung Chung to self-care and development. In response to the poor eating habits identified among the Trekkers families, a series of nutrition workshops incorporating short talks and sharing of healthy recipes was delivered as part of a health empowerment programme. The parents acquired knowledge and skills in healthy eating and cooking in the workshops, and were encouraged to prepare balanced meals and make food choices with nutritional quality for their families. Although there was improvement in dietary knowledge, little change in eating habits was noted in the families after the workshops. There is a need for an in-depth exploration on the barriers and facilitators that low-income families encounter in helping their adolescent children adopt and sustain a healthy eating habit.

Although personal factors of dietary habit among children have been well investigated, whether the parents and adolescents from low income families know, believe or act to tackle the barriers is unknown. Most observational and qualitative studies only identified family correlates of children's eating habit, but did not elaborate on how the families address these factors. A few studies have explored the parent-reported strategies on children's eating habit in western countries, but it is not known whether they are applicable to Hong Kong families whose dietary culture, social environment and family structure are different. Besides, perception difference of family determinants between adolescents and parents is also highlighted in family research. Adolescents tend to focus on personal and social factors such as food preference and personal health benefits, while parents provide additional insight in family food preparation and dietary pattern. Therefore, understanding the barriers, facilitators and strategies to adopt healthy eating habit from both parents and adolescents is crucial for intervention planning in local context.

The investigators propose to use the Knowledge, Attitude and Practice (KAP) explanatory model to explore whether an individual knows, believes, and practices healthy eating. This study will identify the "knowledge of dietary recommendation and health benefits/harms of selected food groups; attitudes in believing, accepting and complying to dietary recommendations for health benefits; and practices of healthy eating" among the families. With the enablers and barriers addressed by KAP model, respective approaches to enhance the adoption of healthy eating behaviors will be explored. These will formulate a framework of the family factors with strategies corresponding to the KAP among the parents and adolescents from low-income families. The investigators will collect data from parent-adolescent pairs to complement information from previous research that collected data from a single source.

Aims:

To investigate the barriers, facilitators and strategies that enable adolescents from low income families to develop a healthy eating habit. The objectives are:

1. To identify the knowledge, attitudes and practices of healthy eating among adolescents
2. To identify individual and family barriers and facilitators of healthy eating in adolescents
3. To explore potential strategies for overcoming corresponding barriers and enforcing facilitators of healthy eating in adolescents

Hypotheses:

1. The attitude of parents from low-income families is the main problem resulted in lack of motivation to encourage healthy dietary behaviors for their adolescents.
2. Food availability at home, food cost and time constraint are the main barriers that hinder healthy eating of adolescents, while perceived health benefit, family meal and parental guidance can enable the healthy eating habit of adolescents.
3. Strategies adopted by low-income family focus on resolving economic and time concern i.e. affordable and time-saving food-related behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Family with an adolescent aged 10-19 by 31 December 2019
* At least one adolescent from the family had completed dietary intake survey on or before 31 December 2019
* Both parent and child have given written consent

Exclusion Criteria:

* Parent or child cannot speak Cantonese
* Neither parent is the primary caregiver of the child

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: They will be sampled from families of the TFES with self-reported dietary habit survey completed by the adolescent (aged 10-19 years). Purposeful sampling of an equal number of families whose adolescents have self-reported healthy or unhealthy diets.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Knowledge of healthy eating | Through study completion, an average of 9 months
  * Guided by semi-structured interview guide
  * Questions will cover knowledge of dietary recommendation, health benefits/ harms, food choice and access to selected food categories
Attitude of healthy eating | Through study completion, an average of 9 months
  * Guided by semi-structured interview guide
  * Questions will cover attitudes in believing, accepting and complying to dietary recommendation for health benefits
Eating behaviours | Through study completion, an average of 9 months
  * Guided by semi-structured interview guide
  * Questions will cover practices of personal and family eating behaviors, including home food environment, family cooking/ meals and parental guidance

SECONDARY OUTCOMES:
Barriers of healthy eating | Through study completion, an average of 9 months
  * Guided by semi-structured interview guide
  * Follow-up questions will cover the barriers encountered based on dietary KAP
Facilitators of healthy eating | Through study completion, an average of 9 months
  * Guided by semi-structured interview guide
  * Follow-up questions will cover the facilitators encountered based on dietary KAP
Strategies for healthy eating | Through study completion, an average of 9 months
  * Guided by semi-structured interview guide
  * Follow-up questions will cover potential strategies for resolving the barriers and promoting facilitators of healthy eating

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Lo Kuen Lam, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided